CLINICAL TRIAL: NCT04615091
Title: "Prognostic Role of Portal Hypertension Assessed by Non-invasive Methods to Stratify Surgical Risk in Compensated Advanced Chronic Liver Disease Patients Undergoing Elective Extrahepatic Surgery: ELASTOSURGERY STUDY."
Brief Title: Non-invasive Methods and Surgical Risk Stratification in Cirrhotics Undergoing Elective Extrahepatic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Antonio Colecchia, Chair Gastroenterology Unit A, Borgo Trento, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: 39512
Record Dates: First submitted 2020-09-18; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Advanced Chronic Liver Disease; Surgery--Complications
Keywords: liver stiffness; spleen stiffness; portal hypertension; liver cirrhosis; extrahepatic surgery; transient elastography; fibroscan
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ELASTO-SURGERY study aims to evaluate the prognostic role of portal hypertension evaluated by non-invasive methods in predicting post-operative morbidity (at 90 days) and mortality (at 365 days) in patients with advanced chronic liver disease undergoing elective extrahepatic surgery.

DETAILED DESCRIPTION:
In the last years, the life expectancy of ACLD patients has increased due to the improvement of the therapeutic strategies of the complications of cirrhosis. .Although surgical procedures have become less invasive the mortality rate in ACLD patients undergoing extrahepatic surgery remains high. For these reasons, an accurate prediction of operative risk for patient-tailored surgical planning becomes crucial.

Purpose of the study: To evaluate the prognostic role of portal hypertension by non- invasive methods in predicting post-operative complications in ACLD patients undergoing elective extrahepatic surgery.

Study type: An international multicenter, prospective, uncontrolled observational study

Study design: In cirrhotic patients undergoing extrahepatic surgery, within one month, a complete baseline evaluation is provided. Baseline evaluation (T0) includes: signature of informed consent, clinical history of liver disease, comorbidities and risk factors for hepato-biliary complications; complete laboratory tests; liver and spleen elastography (with Transient Elastography, ARFI or 2D-SWE).

After surgery, each patient is evaluated at T1 (+90 days) with Elastography, laboratory tests, clinical examination and T2 (+ 365 days) by a clinical examination.

Each center will prospectively collect data according to an electronic e-CFR on REDCap (Research Electronic Data Capture) system, a web application designed to support data capture for research studies in a secure manner.

Study duration: The study period will last approx. 730 days, with a planned follow-up of 365 days after surgical intervention

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs;
* Advanced chronic liver disease (LSM>10 kPa)
* Any etiology (viral, metabolic, alcoholic, cholestatic and autoimmune);
* Elective extrahepatic surgery planned within three months and requiring regional or general anaesthesia;
* Patients are willing and able to give informed consent

Exclusion Criteria:

* Presence of hepatic decompensation at the time of informed consent or previous events of hepatic decompensation during the last three months before enrollment.
* Presence of portal vein thrombosis
* Previous placement of TIPS,
* Prior liver transplantation,
* Surgical resection or shunt.
* Presence of active HCC that needed treatment at the time of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced chronic liver disease patients who are planned an elective extrahepatic surgery (abdominal, orthopaedics and thoracic-cardiovascular surgeries)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Early post-surgical (at +90 days) complications after extrahepatic surgery | 90 days after surgery
  Complications related to the surgical procedure and/or liver disease after the extrahepatic elective surgery

SECONDARY OUTCOMES:
The liver-related events and overall survival at +90 days and + 360 days after extrahepatic surgery | 360 days after surgery
  Liver-related events (decompensation, TIPS placement, liver transplantation) or death (liver e non-liver related) at 90 days 360 days from the elective extra-hepatic surgery

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO COLECCHIA, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; DAVIDE FESTI, MD, Study Chair — University of Bologna; GIOVANNI MARASCO, MD; PhD, Study Chair — University of Bologna; CATERINA CUSUMANO, MD, Study Chair — Azienda Ospedaliera Universitaria Integrata Verona; KAMELA GJINI, Study Chair — Azienda Ospedaliera Universitaria Integrata Verona; FEDERICO RAVAIOLI, MD, Study Chair — University of Bologna; ELTON DAJTI, MD, Study Chair — University of Bologna
Locations (37):
- Yale New Haven Hospital, New Haven, Connecticut, United States
- Medical University of Vienna, Vienna, Austria
- Canada (2):
  - University of Alberta Hospital, Edmonton
  - McGill University Health Centre, Montreal
- Odense University Hospital, Odense, Denmark
- France (10):
  - University hospital of Angers, Angers
  - Hopital Jean Verdier, Bondy
  - Hôpital Jean Verdier, Bondy
  - Bordeaux University Hospital, Bordeau
  - Hôpital Beaujon, Clichy
  - Hospices Civils de Lyon Hopital Hotel Dieu, Lyon
  - Centre Hospitalier de Montpellier, Montpellier
  - hôpital Antoine-Béclère, Hôpitaux Universitaires Paris-Sud, Assistance Publique-Hôpitaux de Paris, Paris
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Purpan Hospital Toulouse, Toulouse
- University Hospital Leipzig, Leipzig, Germany
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- Italy (11):
  - Aoui Borgo Trento, Verona, VR
  - Clinica di Gastroenterologia ed Epatologia Ancona, Ancona
  - Gastroenterology Unit - Azienda Ospedaliera Universitaria Sant'Orsola - Malpighi, Bologna
  - Ospedale di Bolzano, Bolzano
  - Azienda ospedaliero-universitaria Careggi, Florence
  - Policlinico di Milano, Milan
  - Policlinico di Modena, Modena
  - Gastroenterology Unit, University of Palermo, Palermo
  - Università Sapienza, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - ASUGI Clinica Patologie del Fegato, Clinica Chirurgica, Trieste
- South Korea (3):
  - Hanyang University Guri Hospital, Hanyang
  - Boramae Internal Medicine, Seoul
  - Yonsei University College of Medicine, Seoul
- Spain (2):
  - Barcelona Hepatic Hemodynamic Lab. Liver Unit. Hospital Clinic. Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
- Switzerland (2):
  - Inselspital, Bern
  - Ente Ospedaliero Cantonale, Lugano
- United Kingdom (2):
  - UCL Sheila Sherlock, London
  - Room Nottingham Digestive Diseases Centre BRU, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uyei J, Taddei TH, Kaplan DE, Chapko M, Stevens ER, Braithwaite RS. Setting ambitious targets for surveillance and treatment rates among patients with hepatitis C related cirrhosis impacts the cost-effectiveness of hepatocellular cancer surveillance and substantially increases life expectancy: A modeling study. PLoS One. 2019 Aug 26;14(8):e0221614. doi: 10.1371/journal.pone.0221614. eCollection 2019. PMID 31449554
- [Background] Newman KL, Johnson KM, Cornia PB, Wu P, Itani K, Ioannou GN. Perioperative Evaluation and Management of Patients With Cirrhosis: Risk Assessment, Surgical Outcomes, and Future Directions. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2398-2414.e3. doi: 10.1016/j.cgh.2019.07.051. Epub 2019 Jul 31. PMID 31376494
- [Background] Reverter E, Cirera I, Albillos A, Debernardi-Venon W, Abraldes JG, Llop E, Flores A, Martinez-Palli G, Blasi A, Martinez J, Turon F, Garcia-Valdecasas JC, Berzigotti A, de Lacy AM, Fuster J, Hernandez-Gea V, Bosch J, Garcia-Pagan JC. The prognostic role of hepatic venous pressure gradient in cirrhotic patients undergoing elective extrahepatic surgery. J Hepatol. 2019 Nov;71(5):942-950. doi: 10.1016/j.jhep.2019.07.007. Epub 2019 Jul 19. PMID 31330170
- [Background] Colecchia A, Ravaioli F, Marasco G, Colli A, Dajti E, Di Biase AR, Bacchi Reggiani ML, Berzigotti A, Pinzani M, Festi D. A combined model based on spleen stiffness measurement and Baveno VI criteria to rule out high-risk varices in advanced chronic liver disease. J Hepatol. 2018 Aug;69(2):308-317. doi: 10.1016/j.jhep.2018.04.023. Epub 2018 May 3. PMID 29729368
- [Background] Colecchia A, Montrone L, Scaioli E, Bacchi-Reggiani ML, Colli A, Casazza G, Schiumerini R, Turco L, Di Biase AR, Mazzella G, Marzi L, Arena U, Pinzani M, Festi D. Measurement of spleen stiffness to evaluate portal hypertension and the presence of esophageal varices in patients with HCV-related cirrhosis. Gastroenterology. 2012 Sep;143(3):646-654. doi: 10.1053/j.gastro.2012.05.035. Epub 2012 May 27. PMID 22643348
- [Background] Ma X, Wang L, Wu H, Feng Y, Han X, Bu H, Zhu Q. Spleen Stiffness Is Superior to Liver Stiffness for Predicting Esophageal Varices in Chronic Liver Disease: A Meta-Analysis. PLoS One. 2016 Nov 9;11(11):e0165786. doi: 10.1371/journal.pone.0165786. eCollection 2016. PMID 27829057
- [Background] Cescon M, Colecchia A, Cucchetti A, Peri E, Montrone L, Ercolani G, Festi D, Pinna AD. Value of transient elastography measured with FibroScan in predicting the outcome of hepatic resection for hepatocellular carcinoma. Ann Surg. 2012 Nov;256(5):706-12; discussion 712-3. doi: 10.1097/SLA.0b013e3182724ce8. PMID 23095613
- [Background] Marasco G, Colecchia A, Dajti E, Ravaioli F, Cucchetti A, Cescon M, Festi D. Prediction of posthepatectomy liver failure: Role of SSM and LSPS. J Surg Oncol. 2019 Mar;119(3):400-401. doi: 10.1002/jso.25345. Epub 2018 Dec 18. No abstract available. PMID 30561034